CLINICAL TRIAL: NCT02125708
Title: Core-temperature Monitoring in Patients With PPROM for Early Detection of Chorioamnionitis - a Pilot Study
Brief Title: Core-temperature Monitoring in Patients With PPROM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no acitve participants
Sponsor: Medical University of Vienna (Other)
Collaborators: The Obstetrics and Gynaecology Clinic Narodni Front (Other)
Responsible Party: Principal Investigator, Associate Prof. Ljubomir Petricevic MD, Ass. Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0012014
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2016-11

CONDITIONS: Preterm Premature Rupture of Fetal Membranes
Keywords: preterm prelabor rupture of membranes; Ovula Ring; body-core-temperature; biomarkers; Single pregnancies; PPROM; gestation week 22 and 27
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OvulaRing® (Other): Twenty patients with verified PPROM between gestation week 22 and 27 should be included. After gynecological and physical examination within verification of PPROM women will be informed about the study and invited to participate in this study. Subsequently informed consent will be obtained and the OvulaRing® placed into the vaginal fornix.
  Interventions: Device: OvulaRing®

INTERVENTIONS:
Device: OvulaRing® — The OvulaRing® is a non-invasive thermometer measuring the intravaginal temperature every 5 minutes. It was originally invented to assess the moment of ovulation and optimize fertility. This plastic ring including a high-tech-sensor thermometer should be placed into the vaginal fornix for a maximum of 30 days, measuring the intravaginal core-temperature 288 times a day.

SUMMARY:
The most common reason for preterm prelabor rupture of membrane (PPROM) is an ascendance of infection. Moreover PPROM is one of the main risk factors for chorioamnionitis.

PPROM-related morbidity and mortality is higher in the neonate than in the mother, especially in case of intrauterine inflammation. Of note, the most common biomarkers like CRP and leucocytes are not specific for uterine infections and have not been proven useful in these particular cases. Studies in intensive care medicine could show that there is a possible correlation between onset of infection and body-core-temperature.

The OvulaRing® is a non-invasive thermometer measuring the intravaginal temperature every 5 minutes. It was originally invented to assess the moment of ovulation and optimize fertility.

Twenty patients with verified PPROM between gestation week 22 and 27 should be included in this study. After gynecological and physical examination within verification of PPROM women will be informed and invited to participate in this study. Subsequently informed consent will be obtained and the OvulaRing® placed into the vaginal fornix.

The investigators aim to describe a possible correlation between core-temperature and common biomarkers in clinical use for the detection of chorioamnionitis in patients with PPROM to possibly assess the optimal time for delivery subsequently.

DETAILED DESCRIPTION:
Introduction A prelabor rupture of membranes (PROM) is defined as a loss of amniotic fluid within a rupture of amniotic membrane before the onset of labour, as preterm prelabor rupture of membranes (PPROM) refers to PROM before 37+0 weeks of gestation.

PPROM occurs in 3 percent of pregnancies and is associated with one third of preterm births. There are multiple risk-factors for PPROM as maternal physiologic, genetic, and environmental as well as life-style factors. Of note, history of PPROM in a previous pregnancy, antepartum bleeding, cigarette smoking and genital tract infections, as the single most identifiable risk factor, are strongly associated with PPROM.

PPROM is diagnosed by the clinical loss of fluid from the cervical os. In case of not immediately visible amniotic fluid loss during the gynecological inspection, it can be diagnosed by ultrasound and verified by tests like the Amnisure© or the Fertisave© which detect the alpha microgloubulin 1 or the IGF binding protein of the fetal membranes.

Referring to a randomized controlled trial, the majority of pregnancies with PPROM deliver within one week of membrane rupture.

PPROM-related morbidity and mortality, which depends on gestational age, is higher in the neonate than in the mother, especially in case of intrauterine inflammation. Pulmonary hypoplasia, facial and orthopedic deformation can be the cause of prolonged, early PPROMS.

As the incidence of infection is higher at earlier gestational ages, up to one third of women with PPROM develop serious infections, including chorioamnionitis, endometritis and septicemia. Responsible bacterias are enterococcus, staphylococcus or anaerobic species.

The goal of antibiotic prophylaxis/therapy in PPROM is to reduce maternal and neonatal morbidity and mortality. Women should be observed for signs of infection, including maternal temperature, fetal heart rate, uterine contractions, and periodically common clinical infection markers. As the most common biomarkers like CRP and leucocytes are not specific for uterine infections, they have not been proven useful in these particular cases.

Prematurity is the crucial risk to the fetus with PPROM in the absence of complications like infection, before 34 weeks of gestation. Therefore, expectative management of uncomplicated PPROM-pregnancies at this gestational age is routinely used. This includes blood cell and infection monitoring, avoiding vaginal manipulation, antibiotic prophylaxis/treatment and corticosteroids.

After having reached gestational week 34+ induction of labour is routinely performed, without induction of lung maturity. The goal is a quick reaction to a chorioamnionitis with a prompt delivery.

Materials and Methods This study is conducted as a single centre pilot study in patients with PPROM. The study was approved by the local ethics committee of the Medical University of Vienna (IRB number: 1031/2014). Study center is the Department of Obstetrics and Gynecology of the Medical Universitiy of Vienna General Hospital.

Twenty patients with verified PPROM between gestation week 22 and 27 should be included. After gynecological and physical examination within verification of PPROM women will be informed about the study and invited to participate in this study. Subsequently informed consent will be obtained and the OvulaRing® placed into the vaginal fornix.

The OvulaRing® is a non-invasive thermometer measuring the intravaginal temperature every 5 minutes. It was originally invented to assess the moment of ovulation and optimize fertility. This plastic ring including a high-tech-sensored thermometer should be placed into the vaginal fornix for a maximum of 30 days, measuring the intravaginal core-temperature 288 times a day.

As there is no change of common PPROM-therapy, only clinical standard parameters will lead to the termination of pregnancy. Directly before delivery the OvulaRing® will be removed and the sensor-data will be analyzed with a special software.

Hypothesis In this pilot study, the investigators aim to describe a possible correlation between core-temperature and common biomarkers in clinical use for the detection of chorioamnionitis in patients with PPROM to possibly assess the optimal time for delivery.

A correlation between temperature and CRP, leucocytes and IL-6 should be explored. Later on, these facts may be used to optimize the standard procedures for a PPROM.

In some studies there is pointed out that there is a need for new parameters for chorioamnionitis. Maybe temperature monitoring can become such a new biomarker.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy
* verified PPROM
* gestation week 22 to 27
* signed informed consent (ICF)

Exclusion Criteria:

* multiple pregnancy
* Patient's age under 18 years
* Allergy to epoxide resin or ethylene vinyl acetate (EVA)-Copolymer

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Body-core-temperature | 288 times a day from PPROM-verification until delivery
  The OvulaRing® is a non-invasive thermometer measuring the intravaginal temperature every 5 minutes. This plastic ring including a high-tech-sensor thermometer should be placed into the vaginal fornix for a maximum of 30 days, measuring the intravaginal core-temperature 288 times a day.
  As there is no change of common PPROM-therapy, only clinical standard parameters will lead to the termination of pregnancy. Directly before delivery the OvulaRing® will be removed and the sensor-data will be analyzed with a special software.

SECONDARY OUTCOMES:
CRP | once a day from hospitalization due to PPROM until delivery
Interleukine (IL-) 6 | once a day from hospitalization due to PPROM until delivery
white blood cell count | once a day from hospitalization due to PPROM until delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ljubomir Petricevic, Ass. Prof. M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Obstetrics and Gynecology, Medical University of Vienna, Vienna, Austria